CLINICAL TRIAL: NCT03292159
Title: Safety and Effectiveness of Transcutaneous Vagus Nerve Stimulation Therapy to Improve Motor Recovery After Stroke
Brief Title: Transcutaneous Vagus Nerve Stimulation for Motor Recovery After Stroke
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: funding not continued
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana Foundation, Spaulding Rehabilitation Hospital (Unknown)
Responsible Party: Principal Investigator, Judith Schaechter, Assistant Professor, Department of Radiology, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017P000129
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Stroke; Upper Extremity Paresis
Keywords: stroke; vagus nerve stimulation; upper extremity paresis
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RAVANS (Experimental)
  Interventions: Device: Active RAVANS concurrent with arm motor training
- Sham stimulation (Sham Comparator)
  Interventions: Device: Inactive RAVANS concurrent with arm motor training

INTERVENTIONS:
Device: Active RAVANS concurrent with arm motor training — Patient receives non-painful, sensory-level stimulation to the skin of left outer ear, where nerve endings of the auricular branch of the vagus nerve reside, while participating in arm motor training
  Arms: RAVANS
Device: Inactive RAVANS concurrent with arm motor training — Patient does not receive stimulation delivered to the skin of left outer ear while participating in arm motor training
  Arms: Sham stimulation

SUMMARY:
This study will evaluate the safety and effectiveness of Respiratory-gated Auricular Vagal Afferent Nerve Stimulation (RAVANS) for improving motor recovery after stroke. Subacute stroke patients will receive RAVANS or sham stimulation concurrent with arm motor training during 10 intervention sessions occurring daily for 30 minutes over 2 weeks. The safety and improvements in arm motor function after the intervention will be compared in patients receiving RAVANS to those receiving sham stimulation.

DETAILED DESCRIPTION:
This study will evaluate the safety, feasibility and effectiveness of Respiratory-gated Auricular Vagal Afferent Nerve Stimulation (RAVANS) for improving motor recovery after stroke. Subacute stroke patients will be randomized to RAVANS or sham stimulation groups. Patients will receive RAVANS or sham stimulation concurrent with arm motor training during 10 sessions occurring daily for 30 minutes over 2 weeks. Safety will be compared in patients receiving RAVANS to those receiving sham stimulation. Feasibility will be evaluated by recruitment into the study and retention of enrolled patients. Changes in arm motor function will be compared between RAVANS and sham stimulation groups from baseline to immediately after the intervention period and to function at 3-months after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Supratentorial ischemic or hemorrhagic stroke incurred 4-30 days prior;
* Contralesional UL motor impairment defined by NIHSS item 5 score 1 or 2 (scale 0-4);
* Age ≥ 18;
* Able to provide written informed consent.

Exclusion Criteria:

* Implanted electronic device (e.g., pacemaker, neurostimulator);
* Pregnancy;
* Major psychiatric or medical condition that could interfere with study participation;
* Medical condition affecting left ear that could interfere with delivering RAVANS (e.g., wound, infection, malignancy, hypoesthesia);
* Significant pre-existing disability of stroke-affected UL in activities of daily living due to prior stroke or other medical cause defined by Stroke Impact Scale item 7 (SIS-hand) mean score < 4 (scale: 0-5);
* History of seizure during year before stroke or > 1 post-stroke seizure;
* Significant cognitive or language impairment that would interfere with informed consent or study participation;
* Severe dysphagia;
* Bradycardia defined as resting heart rate < 50 bpm;
* Nonsustained ventricular tachycardia;
* Cardiac conduction disorder (i.e., bundle branch block, heart block, long Q-T syndrome);
* History of asystole;
* History of recurrent vaso-vagal syncope;
* Hypotension defined as blood pressure < 90/60 mmHg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Upper extremity motor impairment | Baseline to just after 10 intervention sessions, and baseline to 3 months post-stroke
  Change in upper extremity subtest of Fugl Meyer Assessment (FMA-UE) score

SECONDARY OUTCOMES:
Upper extremity motor function | Baseline to just after 10 intervention sessions, and baseline to 3 months post-stroke
  Change in Action Research Arm Test (ARAT) score
Grip force control | Baseline to just after 10 intervention sessions, and baseline to 3 months post-stroke
  Change in accuracy, variability and temporal structure of performance on a grip force control task
Upper extremity disability | Baseline to 3 months post-stroke
  Change in hand subtest of Stroke Impact Scale (SIS-hand) score
Mood state, anxiety and depression | Baseline to 3 months post-stroke
  Change in Hospital Anxiety and Depression Scale (HADS) scores

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States